CLINICAL TRIAL: NCT04933838
Title: Evaluation of an Effectiveness and Safety of Atelocollagen in the Management of Chronic Non-specific Low Back Pain: A Prospective, Randomized, Comparative Pilot Study
Brief Title: Effectiveness and Safety of Atelocollagen in the Management of Chronic Non-specific Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University (Other)
Responsible Party: Principal Investigator, Jeeyoun Moon, Associate professor, Seoul National University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2011-183-1177
Record Dates: First submitted 2021-06-01; First posted 2021-06-22 (Actual); Last update posted 2022-09-14 (Actual); Status verified 2022-09

CONDITIONS: Low Back Pain
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (Placebo Comparator): 1% licocaine 3 mL + Normal saline 3 mL mixture
  Interventions: Device: atelocollagen
- Atelocollagen group (Experimental): 1% lidocaine 3 mL + atelocollagen 3 mL mixture
  Interventions: Device: atelocollagen

INTERVENTIONS:
Device: atelocollagen — This collagen-contained product is used to supplement tendon, ligament, muscle, and (biological) membrane that is missing or damaged during internal/surgical treatment and surgery.
  Patients with chronic low back pain are randomized after obtaining informed consent for the study.
  Participants are divided into group A (atelocollagen) and group B (control). A physical examination for lumbar pain was performed and evaluated trigger points in multifidus, erector spinae, and quadratus lumborum muscles.
  After physical exam, cross sectional area of each muscle is measured by ultrasound in both gorup.
  Group A will receive atelocollagen mixture (atelocollagen 3 mL + 1% lidocaine 3 mL) and group B will receive local anesthetics only (Normal saline 3 mL + 1% lidocaine 3 mL).
  Each participants will be injected 1 mL of injectate into each muscle on both sides (total 6 mL).

SUMMARY:
The purpose of this study was to evaluate the effectiveness and safety of atelocollagen in the management of chronic low back pain with sarcopenia due to degenerative changes.

DETAILED DESCRIPTION:
Patients with chronic low back pain are enrolled and divided into group A (atelocollagen) and group B (control) through randomization after obtaining informed consent.

Investigators record tender points for the multifidus, erector spinae, and quadratus lumborum muscles by physical examination.

Investigators evaluate each muscle using ultrasound according to the assignment of each group, and apply atelocollagen mixture (atelocollagen 3 mL + 1% lidocaine 3 mL) or local anesthetics only (normal saline 3 mL + 1% lidocaine 3 mL) to each muscle on both sides.

The subject of the study performs a total of 3 injections at intervals of 2 weeks, and each measurement variable is collected by visiting 4 weeks and 12 weeks after the last injection.

Changing medications or additive interventions are not allowed before 4 weeks after last injection. Only acetaminophen is allowed as a rescue drug.

ELIGIBILITY:
Inclusion Criteria:

- Non-specific low back pain with persistent paraspinal tenderness of NRS 4 or higher despite conservative treatment (including physical therapy, exercise therapy, oral drug administration, and epidural block) for at least 3 months.

Adults 19 years of age or older

Exclusion Criteria:

- Systemic or local infection Coagulopathy Patients whose structure is difficult to confirm on ultrasound due to significant deformity of the lumbar spine Neoplasm of spine Cognitive disorder Patients with hypersensitivity to local anesthetics or amide-based local anesthetics Patients those who are allergic to or sensitive to atelocollagen ingredients or pork Women who are pregnant, lactating, or planning to become pregnant during the clinical period, or women of childbearing age who are not using available contraceptive methods Those who participated in other clinical trials within 30 days prior to screening or 5 times the half-life of the investigational drug in the clinical trial in which they participated, whichever is longer, whichever is longer Patients with serious systemic diseases

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2021-07-01 (Actual); Primary Completion 2022-03-03 (Actual); Study Completion 2022-04-27 (Actual)

PRIMARY OUTCOMES:
Pain changes in low back pain | 4 weeks after last intervention
  The changes of the 11-point Numeric Rating Scale(NRS) pain score (numeric scale ranges from '0' representing one pain extreme (e.g. "no pain") to '10' representing the other pain extreme (e.g. "pain as bad as you can imagine" or "worst pain imaginable")) after intervention between two groups.

SECONDARY OUTCOMES:
Pain changes in low back pain | 12 weeks after last intervention
  The changes of the 11-point Numeric Rating Scale(NRS) pain score (numeric scale ranges from '0' representing one pain extreme (e.g. "no pain") to '10' representing the other pain extreme (e.g. "pain as bad as you can i
Cross-sectional area | 4, 12 weeks after last intervention
  The changes of cross-sectional area using ultrasound after intervention between two groups.
Oswestry Disability Index(ODI) score | 4, 12 weeks after last intervention
  The changes of ODI score after intervention between two groups.
Satisfaction (participants) | 4 weeks after first intervention
  5-pointed satisfaction scale of intervention (participants)
Satisfaction (pain physician) | 4 weeks after first intervention
  5-pointed satisfaction scale of intervention (pain physician)
Pain related to intervention | 4 weeks after first intervention
  The 11-point Numeric Rating Scale(NRS) pain score (numeric scale ranges from '0' representing one pain extreme (e.g. "no pain") to '10' representing the other pain extreme (e.g. "pain as bad as you can imagine" or "worst pain imaginable")) related to intervention
Medication | 12 weeks after last intervention
  The changes in medication

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Seoul, South Korea